CLINICAL TRIAL: NCT00016068
Title: A Phase III Multicenter Study Of Valganciclovir For The Prevention Of Late Cytomegalovirus Infection After Allogeneic Hematopoietic Stem Cell Transplantation
Brief Title: Valganciclovir to Prevent Cytomegalovirus Infection in Patients Following Donor Stem Cell Transplantation
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Fred Hutchinson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Allocation: Randomized | Masking: Double | Purpose: Supportive Care
Other Study IDs: 1577.00; FHCRC-1577.00; MSKCC-01127; NCI-H01-0072
Record Dates: First submitted 2001-05-06; First posted 2003-01-27 (Estimated); Last update posted 2010-05-17 (Estimated); Status verified 2010-05

CONDITIONS: Infection
Keywords: infection
MeSH Terms: conditions — Infections | interventions — Ganciclovir; Valganciclovir

INTERVENTIONS:
Drug: ganciclovir
Drug: valganciclovir

SUMMARY:
RATIONALE: Antivirals such as valganciclovir act against viruses and may be effective in preventing cytomegalovirus. It is not yet known if valganciclovir is effective in preventing cytomegalovirus.

PURPOSE: This randomized phase III trial is studying valganciclovir to see how well it works in preventing cytomegalovirus in patients who have undergone donor stem cell transplantation.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Compare cytomegalovirus (CMV) disease and non-CMV invasive infection-free survival in patients undergoing allogeneic hematopoietic stem cell transplantation treated with valganciclovir vs placebo.
* Compare the incidence of CMV disease in patients treated with these drugs.
* Compare the incidence of other severe invasive bacterial and fungal infections and overall survival in patients treated with these drugs.

Secondary

* Compare the incidence of CMV infection or disease at baseline and at days 270 and 640 after allogeneic hematopoietic stem cell transplantation in patients treated with these drugs.
* Compare the incidence of herpes simplex virus and varicella-zoster virus infections at baseline and day 270 in patients treated with these drugs.
* Determine the safety of valganciclovir in these patients.
* Compare the quality of life of patients treated with these drugs.
* Compare CMV-specific immune reconstitution in patients treated with these drugs.

OUTLINE: This is a randomized, double-blind, placebo-controlled, multicenter study. Patients are stratified according to participating center, prior neutropenia (yes vs no), and presence of refractory graft-versus-host disease requiring secondary therapy (yes vs no). Patients are randomized to 1 of 2 treatment arms.

* Arm I: Patients receive oral valganciclovir daily.
* Arm II: Patients receive oral placebo daily. Treatment begins around day 80-120 post-transplantation and continues until day 270 post-transplantation in the absence of active infection or unacceptable toxicity. Patients developing active cytomegalovirus (CMV) infection receive induction doses of ganciclovir IV or open-label oral valganciclovir for 1 week followed by open-label oral valganciclovir maintenance dosing until CMV can no longer be detected.

Quality of life is assessed at baseline and days 180 and 270 post-transplantation.

Patients are followed at days 400, 520, and 640 post-transplantation.

PROJECTED ACCRUAL: A total of 184 patients (92 per treatment arm) will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Have undergone allogeneic peripheral blood stem cell, cord blood, or marrow transplantation (related or unrelated, T-cell depleted or non-T-cell depleted, CD34-selected or non-selected, or myeloablative or non-myeloablative) within the past 80-120 days
* Positive pre-transplantation cytomegalovirus (CMV) serology of recipient and/or donor

  * Seropositive recipients with one of the following:

    * CMV infection before day 80, as determined by:

      * pp65 antigenemia
      * CMV DNA in plasma
      * Peripheral blood leukocytes (PBL) or whole blood at any level detected by polymerase chain reaction or hybrid capture
      * CMV pp67 mRNA
      * CMV viremia by blood culture
      * Surveillance bronchoalveolar lavage (culture or cytology)
    * CMV disease more than 6 weeks prior to enrollment
    * Presence of graft-versus-host disease (GVHD) at enrollment

      * Acute GVHD that requires treatment with systemic corticosteroids of doses greater than 0.5 mg/kg OR
      * Chronic clinically extensive GVHD requiring treatment with corticosteroids
    * Continuous prophylaxis with ganciclovir, foscarnet, or cidofovir between engraftment and day 80 OR
  * Seronegative recipient with seropositive donor who has CMV infection before day 80
* No rising or uncontrolled CMV load (pp65 antigenemia levels no greater than 1/slide or no greater than 100 copies of CMV DNA per mL of plasma or per million PBL allowed)
* No CMV disease within 6 weeks prior to randomization
* No leukemic relapse

  * Cytogenetic or molecular relapse allowed

PATIENT CHARACTERISTICS:

Age:

* 16 and over

Performance status:

* Not specified

Life expectancy:

* At least 2 weeks

Hematopoietic:

* Absolute neutrophil count at least 1,000/mm^3 for at least 1 week prior to enrollment

Hepatic:

* Not specified

Renal:

* Creatinine no greater than 2.5 mg/mL

Other:

* No hypersensitivity to ganciclovir or valganciclovir
* No uncontrolled diarrhea or severe gastrointestinal disease that would preclude oral medication
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception during and for 90 days after study participation
* HIV negative
* Proficient in English

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* See Disease Characteristics

Chemotherapy:

* Not specified

Endocrine therapy:

* See Disease Characteristics

Radiotherapy:

* Not specified

Surgery:

* Not specified

Other:

* Prior ganciclovir, foscarnet, cidofovir, high-dose acyclovir, or valacyclovir as prophylaxis or preemptive therapy allowed
* No concurrent prophylactic foscarnet, cidofovir, or ganciclovir (IV or oral)
* No concurrent prophylactic high-dose acyclovir (more than 800 mg twice daily), valacyclovir (more than 500 mg twice daily), cidofovir (more than 0.5 mg/kg per week), or famciclovir (more than 500 mg/day) except for limited treatment courses at higher doses for varicella-zoster virus infections

  * Concurrent low-dose (≤ 0.5 mg/kg per week) cidofovir allowed for limited treatment courses

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 184 (Estimated)
Dates: Start 2001-01; Study Completion 2007-09 (Actual)

PRIMARY OUTCOMES:
Late cytomegalovirus infection by plasma PCR positivity

CONTACTS AND LOCATIONS:
Overall Officials: Michael Boeckh, MD, Study Chair — Fred Hutchinson Cancer Center
Locations (7):
- United States (7):
  - City of Hope Comprehensive Cancer Center, Duarte, California
  - University of Florida Shands Cancer Center, Gainesville, Florida
  - Barbara Ann Karmanos Cancer Institute, Detroit, Michigan
  - Mayo Clinic Cancer Center, Rochester, Minnesota
  - Memorial Sloan-Kettering Cancer Center, New York, New York
  - M.D. Anderson Cancer Center at University of Texas, Houston, Texas
  - Fred Hutchinson Cancer Research Center, Seattle, Washington

REFERENCES:
- [Derived] Boeckh M, Nichols WG, Chemaly RF, Papanicolaou GA, Wingard JR, Xie H, Syrjala KL, Flowers ME, Stevens-Ayers T, Jerome KR, Leisenring W. Valganciclovir for the prevention of complications of late cytomegalovirus infection after allogeneic hematopoietic cell transplantation: a randomized trial. Ann Intern Med. 2015 Jan 6;162(1):1-10. doi: 10.7326/M13-2729. PMID 25560711